CLINICAL TRIAL: NCT04369001
Title: Program ACTIVE: Implementing a Cognitive Behavioral Therapy and Physical Activity Program for Black Men With Comorbid Diabetes and Depression
Brief Title: Program ACTIVE: Phase 2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to covid-19 and social distancing, this study was terminated.
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jaclynn Hawkins, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ProgramACTIVE; P30DK092926 (NIH)
Record Dates: First submitted 2020-04-14; First posted 2020-04-30 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 2; Depression
Keywords: Type 2 diabetes; Depression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): (Program ACTIVE n=20) Participants randomized into the Program ACTIVE group will receive a gym membership to a local, Detroit-based community recreation facility where they will complete 150 minutes of exercise per week for 12 weeks and will receive 10 sessions (once weekly) of CBT therapy sessions. Exercise per week will be documented using exercise logs. Exercise logs will be given to research staff at the end of the 12-week timeframe; all exercise logs will be kept organized respective to the participant identification number and related documents (questionnaires and surveys). To ensure treatment fidelity, three CBT and three physical activity sessions will be selected at random and recorded and rated for fidelity to the above content by our research team.
  Interventions: Behavioral: Community-Based Exercise; Behavioral: Cognitive Behavioral Therapy
- Enhanced Usual Care (No Intervention): (EUC n=20) Participants randomized to enhanced usual care will receive referrals to community mental health providers, pedometers, gym memberships to a community-based venue, and intervention patient manuals. Participants will not be required to report any use of resources offered or change their course of treatment in any way. Based on several years of experience in Detroit, providing all participants with referrals, pedometers, gym access and educational materials minimizes ethical concerns regarding assignment of underserved populations to receive a no-treatment control.

INTERVENTIONS:
Behavioral: Community-Based Exercise — Participants will complete 150 minutes of exercise per week for 12 weeks. Exercise per week will be documented using exercise logs. The exercise protocol will be a culturally-tailored community-based exercise intervention based on the aerobic exercise goals used in the Program ACTIVE study and psychoeducational materials adapted from Program ACTIVE based on feedback from Black men with T2D. Exercise in Program ACTIVE will be obtained through individualized community-based activities that participants in the focus groups indicate as feasible rather than the highly controlled laboratory environment. Exercise goals will be adapted to accommodate the physical and medical restrictions of an older-adult diabetes population.
  Other Names: EXER
  Arms: Intervention Group
Behavioral: Cognitive Behavioral Therapy — Participants will receive 10 sessions of CBT using a manualized approach based on Beck's model of cognitive therapy. Sessions are to be completed once weekly in conjunction with weekly exercise. The Program ACTIVE CBT intervention includes: presentation of CBT model; thought records, cognitive distortions, counterarguments, cognitive reframing, automatic thoughts, core beliefs, and relapse prevention. Session goals will be tailored to the needs of men so that the order of topics may vary. Each session will begin with the designation of session goals, review of previously assigned homework, and introduction of new concepts and skills. Individually-tailored homework assignments designed to provide practice with the concepts/skills of the session will be assigned.
  Other Names: CBT
  Arms: Intervention Group

SUMMARY:
The present study seeks to tailor the original Program ACTIVE (Adults Coming Together to Increase Vital Exercise) to meet the cultural norms and needs of adult Black men with comorbid Type 2 diabetes and depression by using focus groups comprised of Black men with Type 2 diabetes. The use of peer perspectives allows for an improved strategy to reach, retain, and improve outcomes in this population.

Following the tailoring of program materials, the intervention (Program ACTIVE) will be facilitated with Black men with comorbid Type 2 diabetes and depression using evidence-based cognitive behavioral therapy and community-based exercise interventions.

DETAILED DESCRIPTION:
Black men have a 1.5 higher incidence of type 2 diabetes (T2D) compared to non-Hispanic White men and are twice as likely to die from diabetes-related complications. Additionally, Black men are more likely to be diagnosed with T2D compared to non-Hispanic White men, and this disparity increases among men over the age of 55. Poor diabetes self-management dramatically increases the risk for micro and macrovascular complications. Because Black men have worsened glycemic management compared to non-Hispanic White men, their risk for these diabetes complications is higher. In addition to physical complications, patients with T2D are twice as likely to experience depressive symptoms than those without T2D. Depressive symptoms are associated with suboptimal blood glucose levels and diabetes complications. A growing body of literature also demonstrates the critical role of gender in the management of physical and mental health conditions, including T2D and depression, and shows that male gender norms may conflict with help-seeking and healthy behaviors.

Program ACTIVE (Adults Coming Together to Increase Vital Exercise) is an evidence-based, cognitive behavioral therapy (CBT) and community-based exercise (EXER) intervention that aims to improve diabetes and depression outcomes that was developed for adults with type 2 diabetes. Research suggests that Black men have more adverse life experiences than men of other racial/ethnic groups, and consequently, experience worsened mental health. Since CBT and exercise programs are the gold standard for treating comorbid T2D and depression, tailoring these existing interventions to meet the needs of Black men with T2D is critical, especially given that high rates of T2D and depression exist in low income Black communities. Additionally, there is a dearth of literature about barriers and facilitators to mental health care utilization and exercise among Black men with T2D. The proposed study seeks to:

Aim 1 (Pre-implementation): Adapt an evidence-based intervention to work with Black men with T2D and depression in a community-based clinic. Adaptation and refinement, guided by the TDF domains, will involve:

1. conducting focus groups with Black men with comorbid T2D and depression to assess barriers and facilitators to mental health care utilization and exercise and to evaluate feasibility and acceptability of intervention materials.

Aim 2: Assess the impact of the implementation intervention strategies developed in Aim 1 by:

1. conducting a pilot randomized controlled trial of Program ACTIVE to evaluate participant recruitment and retention rates, treatment and intervention satisfaction and estimate intervention effect sizes on our primary outcomes of glycemic control (HbA1c) and depression as well as on secondary outcomes such as self-management behaviors and diabetes social support at baseline, 3 and 6 months post-intervention. Data from the pilot trial will help refine recruitment strategies, training materials, and the implementation protocol to be used in a larger pilot trial.
2. conducting qualitative interviews, guided by the TDF domains, to better understand the acceptability and sustainability of M-Action as routine practice in a community-based clinic.

ELIGIBILITY:
Inclusion Criteria: (must include all of the following):

* age 18 or older
* male sex assigned at birth
* Black
* a diagnosis of T2D for one year duration or longer
* ambulatory status
* major depression lasting 2 weeks or longer with no current evidence of psychotic symptoms. All persons scoring >5 on a PHQ-9 administered via a telephone screening (administered by a research assistant or project coordinator) will be invited to participate. Patients who are currently prescribed antidepressant medications for 6 weeks or longer and who meet diagnostic criteria for major depression without psychotic features will be included. Patients who are currently receiving only medication management from a psychiatrist will be included. Respondents who meet eligibility criteria will be invited to participate in the baseline screening assessment.

Exclusion Criteria:

* Stage 2 hypertension as defined by JNC VIII
* recent cardiac events
* recent laser surgery for proliferative retinopathy
* history of stroke
* lower limb amputation
* asensory peripheral neuropathy
* aortic stenosis or other severe valvular heart disease
* atrial fibrillation
* severe COPD (e.g., basal oxygen)
* class III or IV heart failure or medical instability
* Patients who report the use of a current antidepressant medication for 5 weeks or less will be excluded or deferred for later screening after the 6-week period. Patients who are currently receiving psychotherapy services from a mental health provider will be excluded. Psychiatric exclusion criteria include: active suicidal ideation or a history of a suicide attempt, bipolar depression or history of psychotic disorder, current substance use or dependent disorder.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligible participants must identify as male-assigned at birth and currently identify as a man.
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change of Metabolic Control | HbA1c will be collected once at baseline, once immediately after the completion of the exercise and behavioral interventions, 3-month post treatment assessment, and 6-months post treatment assessment.
  Metabolic Control will be measured via hemoglobin A1c (HbA1c). HbA1c will be collected using the DCA 2000 point-of-care testing instrument.
Change of Depression Scores | Depression scores will be collected once at baseline, once immediately after the completion of the exercise and behavioral interventions, 3-month post treatment assessment, and 6-months post-treatment assessment.
  Depression will be measured using the PHQ-9 (score >=10) and The BDI-II, a 21-item self-administered questionnaire used to assess symptoms of depression. Depression will be measured using the Beck Depression Inventory (BDI-II). BDI-II items have been designed to correspond with DSM-IVTR diagnostic criteria. The BDI-II has been shown to have excellent test-retest reliability and validity when used in general populations as well for use with diabetes samples.

SECONDARY OUTCOMES:
Change of Regimen Adherence | Perceived Diabetes Self-Management scores will be collected once at baseline, once immediately after the completion of the exercise and behavioral interventions, 3-month post treatment assessment, and 6-months post-treatment assessment.
  Regimen adherence will be measured using the Perceived Diabetes Self-Management Scale, a self-report questionnaire used to measure a broad range of management behaviors, such as insulin management, dietary management, blood glucose monitoring, symptom response, and parent assistance/supervision. The responses for the PDSMS items range from 1 = "Strongly Disagree" to 5 = "Strongly Agree." Four of the items (#s 1, 2, 6, & 7) are worded such that high agreement signifies low self-efficacy or perceived competence. These four items are reverse scored prior to being added to the other four items. The total PDSMS score can range from 8 to 40, with higher scores indicating more confidence in self-managing one's diabetes.
Change of Adherence to Gender Norms | Male Role Norms Inventory-Short Form scores will be collected once at baseline, once immediately after the completion of the exercise and behavioral interventions, 3-month post treatment assessment, and 6-months post-treatment assessment.
  Adherence to gender norms will be measured using the Male Role Norms Inventory-Short Form. The items are separated into seven subscales: Restrictive Emotionality, Self-Reliance Through Mechanical Skills, Negativity Toward Sexual Minorities, Avoidance of Femininity, Importance of Sex, Toughness, and Dominance. Response Options are on a 7-point scale ranging from strongly disagree = 1 to strongly agree = 7. Higher scores indicate more traditional gender role beliefs.
Change of Body Mass Index | Body Mass Index will be collected once at baseline, once immediately after the completion of the exercise and behavioral interventions, 3-month post treatment assessment, and 6-months post-treatment assessment.
  Body Mass Index will be calculated using height and weight. Height will be measured using a stadiometer.
Change of Weight | Weight will be collected once at baseline, once immediately after the completion of the exercise and behavioral interventions, 3-month post treatment assessment, and 6-months post-treatment assessment.
  Weight will be measured on a high quality, calibrated digital scale.
Change of Blood Pressure | Blood Pressure will be collected once at baseline, once immediately after the completion of the exercise and behavioral interventions, 3-month post treatment assessment, and 6-months post-treatment assessment.
  Blood Pressure will be measured using the auscultatory method assessing for both diastolic and systolic pressure.
Change of Diabetes Social Support | Diabetes Social Support scores will be collected once at baseline, once immediately after the completion of the exercise and behavioral interventions, 3-month post treatment assessment, and 6-months post-treatment assessment.
  Diabetes Social Support will be measured using the Diabetes Social Support Questionnaire. The questionnaire is a 5-item survey with answers ranging from 1 - "I receive none" to 5 - "I don't need help." Total scores range from a minimum of 5, indicating low social support for diabetes treatment and management, to 25, a high indication of social support for diabetes treatment and management.
Change of Diabetes-Related Distress | Diabetes Related Distress scores will be collected once at baseline, once immediately after the completion of the exercise and behavioral interventions, 3-month post treatment assessment, and 6-months post-treatment assessment.
  Diabetes-related Distress will be measured using Diabetes Distress Scale (Short Form-12). The Diabetes Distress Scale items pertain to common emotions perceived by individuals self-managing their diabetes. The scale, ranging from 1 = not a problem to 6 = very serious problem scores the degree to which the items have distressed the individual.
Change of Diabetes Quality of Life | Diabetes Quality of Life scores will be collected once at baseline, once immediately after the completion of the exercise and behavioral interventions, 3-month post treatment assessment, and 6-months post-treatment assessment.
  Diabetes Quality of Life will be used to measure quality of life. The DQoL measure consists of 46 items ranked on a 5-point Likert scale. Total scores range from 0 (lowest possible QoL) to 100 (highest possible QoL).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Centers for Disease Control and Prevention. Age-Adjusted Percentage of Civilian, Noninstitutionalized Population with Diagnosed Diabetes, by Race and Sex, United States, 1980-2011, 2013. http://www.cdc.gov/diabetes/statistics/prev/national/figraceethsex.htm
- [Background] Centers for Disease Control and Prevention. National Diabetes Statistics Report: Estimates of Diabetes and Its Burden in the United States, 2014. Atlanta, GA: US Department of Health and Human Services, 2014.
- [Background] Egede LE, Mueller M, Echols CL, Gebregziabher M. Longitudinal differences in glycemic control by race/ethnicity among veterans with type 2 diabetes. Med Care. 2010 Jun;48(6):527-33. doi: 10.1097/MLR.0b013e3181d558dc. PMID 20473215
- [Background] Liburd LC, Namageyo-Funa A, Jack L Jr. Understanding "masculinity" and the challenges of managing type-2 diabetes among African-American men. J Natl Med Assoc. 2007 May;99(5):550-2, 554-8. PMID 17534013
- [Background] Seawell AH, Hurt TR, Shirley MC. The Influence of Stress, Gender, and Culture on Type 2 Diabetes Prevention and Management Among Black Men: A Qualitative Analysis. Am J Mens Health. 2016 Mar;10(2):149-56. doi: 10.1177/1557988315580132. Epub 2015 Apr 9. PMID 25862692
- [Background] Hawkins, J, Kieffer EC, Sinco B et al.
- [Background] Hawkins J, Watkins DC, Kieffer E, Spencer M, Piatt G, Nicklett EJ, Lebron A, Espitia N, Palmisano G. An Exploratory Study of the Impact of Gender on Health Behavior Among African American and Latino Men With Type 2 Diabetes. Am J Mens Health. 2017 Mar;11(2):344-356. doi: 10.1177/1557988316681125. Epub 2016 Dec 5. PMID 27923970
- [Background] de Groot M, Doyle T, Kushnick M, Shubrook J, Merrill J, Rabideau E, Schwartz F. Can lifestyle interventions do more than reduce diabetes risk? Treating depression in adults with type 2 diabetes with exercise and cognitive behavioral therapy. Curr Diab Rep. 2012 Apr;12(2):157-66. doi: 10.1007/s11892-012-0261-z. PMID 22350739
- [Background] Holden KB, McGregor BS, Blanks SH, Mahaffey C. Psychosocial, socio-cultural, and environmental influences on mental health help-seeking among African-American men. J Mens Health. 2012 Jun 1;9(2):63-69. doi: 10.1016/j.jomh.2012.03.002. PMID 22905076
- [Background] Watkins DC, Hawkins J, Mitchell JA. The Discipline's Escalating Whisper: Social Work and Black Men's Mental Health. Res Soc Work Pract. 2015 Mar;25(2):240-250. doi: 10.1177/1049731514526621. Epub 2014 Mar 19. PMID 31289430
- [Background] Watkins DC, Jefferson SO. Recommendations for the use of online social support for African American men. Psychol Serv. 2013 Aug;10(3):323-32. doi: 10.1037/a0027904. Epub 2012 Aug 27. PMID 22924797
- [Background] Watkins DC. Depression over the adult life course for African American men: toward a framework for research and practice. Am J Mens Health. 2012 May;6(3):194-210. doi: 10.1177/1557988311424072. Epub 2011 Nov 21. PMID 22105067
- [Background] Williams DR. The health of men: structured inequalities and opportunities. Am J Public Health. 2003 May;93(5):724-31. doi: 10.2105/ajph.93.5.724. PMID 12721133
- [Background] Cane J, O'Connor D, Michie S. Validation of the theoretical domains framework for use in behaviour change and implementation research. Implement Sci. 2012 Apr 24;7:37. doi: 10.1186/1748-5908-7-37. PMID 22530986
- [Background] Michigan Department of Community Health. Michigan Primary Care Transformation Project (MIPCT): Information for Michigan POs/PHOs and Payers 2011.
- [Background] Anderson RJ, Freedland KE, Clouse RE, Lustman PJ. The prevalence of comorbid depression in adults with diabetes: a meta-analysis. Diabetes Care. 2001 Jun;24(6):1069-78. doi: 10.2337/diacare.24.6.1069. PMID 11375373
- [Background] Nefs G, Pouwer F, Denollet J, Pop V. The course of depressive symptoms in primary care patients with type 2 diabetes: results from the Diabetes, Depression, Type D Personality Zuidoost-Brabant (DiaDDZoB) Study. Diabetologia. 2012 Mar;55(3):608-16. doi: 10.1007/s00125-011-2411-2. Epub 2011 Dec 24. PMID 22198261
- [Background] de Groot M, Doyle T, Hockman E, Wheeler C, Pinkerman B, Shubrook J, Gotfried R, Schwartz F. Depression among type 2 diabetes rural Appalachian clinic attendees. Diabetes Care. 2007 Jun;30(6):1602-4. doi: 10.2337/dc06-1599. Epub 2007 Mar 12. No abstract available. PMID 17353505
- [Background] Lustman PJ, Freedland KE, Griffith LS, Clouse RE. Fluoxetine for depression in diabetes: a randomized double-blind placebo-controlled trial. Diabetes Care. 2000 May;23(5):618-23. doi: 10.2337/diacare.23.5.618. PMID 10834419
- [Background] de Groot M, Anderson R, Freedland KE, Clouse RE, Lustman PJ. Association of depression and diabetes complications: a meta-analysis. Psychosom Med. 2001 Jul-Aug;63(4):619-30. doi: 10.1097/00006842-200107000-00015. PMID 11485116
- [Background] Egede LE, Zheng D, Simpson K. Comorbid depression is associated with increased health care use and expenditures in individuals with diabetes. Diabetes Care. 2002 Mar;25(3):464-70. doi: 10.2337/diacare.25.3.464. PMID 11874931
- [Background] Ciechanowski PS, Katon WJ, Russo JE. Depression and diabetes: impact of depressive symptoms on adherence, function, and costs. Arch Intern Med. 2000 Nov 27;160(21):3278-85. doi: 10.1001/archinte.160.21.3278. PMID 11088090
- [Background] Egede LE. Major depression in individuals with chronic medical disorders: prevalence, correlates and association with health resource utilization, lost productivity and functional disability. Gen Hosp Psychiatry. 2007 Sep-Oct;29(5):409-16. doi: 10.1016/j.genhosppsych.2007.06.002. PMID 17888807
- [Background] Katon W, Russo J, Von Korff M, Lin E, Simon G, Bush T, Ludman E, Walker E. Long-term effects of a collaborative care intervention in persistently depressed primary care patients. J Gen Intern Med. 2002 Oct;17(10):741-8. doi: 10.1046/j.1525-1497.2002.11051.x. PMID 12390549
- [Background] Zhang X, Norris SL, Gregg EW, Cheng YJ, Beckles G, Kahn HS. Depressive symptoms and mortality among persons with and without diabetes. Am J Epidemiol. 2005 Apr 1;161(7):652-60. doi: 10.1093/aje/kwi089. PMID 15781954
- [Background] Jaggi LJ, Mezuk B, Watkins DC, Jackson JS. The Relationship between Trauma, Arrest, and Incarceration History among Black Americans: Findings from the National Survey of American Life. Soc Ment Health. 2016 Nov;6(3):187-206. doi: 10.1177/2156869316641730. Epub 2016 Oct 20. PMID 27795871
- [Background] Miller, D. B., & M. D. Bennett. 2011. "Special Issue: Challenges, Disparities and Experiences of African American Males." Research on Social Work Practice 21(3): 265-68. doi:10.1177/1049731510393985.
- [Background] Watkins, D. C., & D. M. Griffith. 2013. "Practical Solutions To Addressing Men's Health Disparities: Guest Editorial." International Journal of Men's Health 12(3): 187-94.
- [Background] Cornish EK, McKissic SA, Dean DAL, Griffith DM. Lessons Learned About Motivation From a Pilot Physical Activity Intervention for African American Men. Health Promot Pract. 2017 Jan;18(1):102-109. doi: 10.1177/1524839915614800. Epub 2016 Jul 10. PMID 26637233
- [Background] Griffith DM, Cornish EK, McKissic SA, Dean DA. Differences in Perceptions of the Food Environment Between African American Men Who Did and Did Not Consume Recommended Levels of Fruits and Vegetables. Health Educ Behav. 2016 Dec;43(6):648-655. doi: 10.1177/1090198115626923. Epub 2016 Mar 1. PMID 26932874
- [Background] Griffith, DM, Thorpe RJ, Wong JY. (Ed); Wester, Stephen R. (Ed). (2016). Men's physical health and health behaviors. APA handbook of men and masculinities., (pp. 709-730). Washington, DC, US: American Psychological Association, xxiv, 799 pp.http://dx.doi.org/10.1037/14594-032
- [Background] Sherman LD, Hawkins JM, Bonner T. An Analysis of the Recruitment and Participation of African American Men in Type 2 Diabetes Self-Management Research: A Review of the Published Literature. Soc Work Public Health. 2017 Jan 2;32(1):38-48. doi: 10.1080/19371918.2016.1188742. Epub 2016 Jul 8. PMID 27392167
- [Background] Beck, A.T., Rush, A.J., Shaw, B.F., Emery, G., Cognitive therapy of depression. 1979, New York, NY: The Guilford Press.
- [Background] Babyak M, Blumenthal JA, Herman S, Khatri P, Doraiswamy M, Moore K, Craighead WE, Baldewicz TT, Krishnan KR. Exercise treatment for major depression: maintenance of therapeutic benefit at 10 months. Psychosom Med. 2000 Sep-Oct;62(5):633-8. doi: 10.1097/00006842-200009000-00006. PMID 11020092
- [Background] Mazzeo RS, Tanaka H. Exercise prescription for the elderly: current recommendations. Sports Med. 2001;31(11):809-18. doi: 10.2165/00007256-200131110-00003. PMID 11583105
- [Background] Levant RF, Hall RJ, Rankin TJ. Male Role Norms Inventory-Short Form (MRNI-SF): development, confirmatory factor analytic investigation of structure, and measurement invariance across gender. J Couns Psychol. 2013 Apr;60(2):228-238. doi: 10.1037/a0031545. Epub 2013 Feb 18. PMID 23421776
- [Background] Broadhead WE, Gehlbach SH, de Gruy FV, Kaplan BH. The Duke-UNC Functional Social Support Questionnaire. Measurement of social support in family medicine patients. Med Care. 1988 Jul;26(7):709-23. doi: 10.1097/00005650-198807000-00006. PMID 3393031
- [Background] Fisher L, Glasgow RE, Mullan JT, Skaff MM, Polonsky WH. Development of a brief diabetes distress screening instrument. Ann Fam Med. 2008 May-Jun;6(3):246-52. doi: 10.1370/afm.842. PMID 18474888
- [Background] Reliability and validity of a diabetes quality-of-life measure for the diabetes control and complications trial (DCCT). The DCCT Research Group. Diabetes Care. 1988 Oct;11(9):725-32. doi: 10.2337/diacare.11.9.725. PMID 3066604
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199

DOCUMENTS (1):
  • Informed Consent Form (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT04369001/ICF_000.pdf